CLINICAL TRIAL: NCT05557695
Title: A Non-interventional, Observational Cohort Study of Chronic Lymphocytic Leukaemia Patients Treated With Acalabrutinib in the First-line Setting Through the UK Early Access Programme: Early Access Programme Outcomes In aCalabrutinib (EPIC).
Brief Title: Observational Study of Acalabrutinib in Patients With Chronic Lymphocytic Leukaemia in the United Kingdom
Acronym: EPIC
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: UKCLL Forum (Unknown)
Responsible Party: Sponsor
Other Study IDs: D8220R00033
Record Dates: First submitted 2022-08-24; First posted 2022-09-28 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia, CLL
Keywords: CLL, real-world evidence, acalabrutinib
MeSH Terms: conditions — Leukemia, B-Cell | interventions — acalabrutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients with chronic lymphocytic leukaemia treated with acalabrutinib in first line
  Interventions: Drug: Acalabrutinib

INTERVENTIONS:
Drug: Acalabrutinib — Acalabrutinib
  Other Names: Calquence

SUMMARY:
This is a retrospective observational research study to describe the characteristics and real-world clinical outcomes of patients with chronic lymphocytic leukaemia receiving acalabrutinib in the United Kingdom (the EPIC study). Physicians treating chronic lymphocytic leukaemia patients with acalabrutinib, where the patients started treatment as part of the acalabrutinib Early Access Programme (EAP), will be invited to recruit patients. Clinical data will be extracted from the patients' clinical records in line with local laws. Data from this study will provide UK-specific real-world data on patients who were started on acalabrutinib as part of the UK acalabrutinib EAP.

DETAILED DESCRIPTION:
1. Primary Objectives:

   a. To estimate real-world progression-free survival in patients with CLL who received acalabrutinib in the first-line.
2. Secondary Objectives:

   1. To estimate real-world overall survival in patients with CLL who received acalabrutinib in the first-line.
   2. To describe real-world response rate to acalabrutinib in patients with CLL who received acalabrutinib in the first-line.
   3. To describe the healthcare resource utilisation in patients with CLL who received acalabrutinib in the first-line.
   4. To describe post-progression treatment patterns in patients with CLL who progressed from first-line acalabrutinib.
   5. To describe real-world clinical progression free survival in patients with CLL who received acalabrutinib in the first-line and progressed during acalabrutinib treatment.
   6. To describe acalabrutinib treatment patterns in patients with CLL who received acalabrutinib in the first-line.
   7. To describe baseline clinical and demographic characteristics in patients with CLL who received acalabrutinib in the first-line.

ELIGIBILITY:
The study population will include treatment-naïve patients with chronic lymphocytic lymphoma (CLL)* who meet the following inclusion criteria:

* Treatment-naïve CLL patients who were initiated on acalabrutinib as part of the UK Early Access Programme
* Received their first dose of acalabrutinib between 1 April 2020 and 1 April 2021
* Patients aged ≥18 years old

  * Note: patients later found to have small lymphocytic lymphoma (SLL) may also be included in the EAP.

Exclusion Criteria:

- None listed in study protocol

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment-naïve adults (≥18 years old) with chronic lymphocytic lymphoma (CLL) who were initiated on acalabrutinib as part of the UK acalabrutiinib early access programme and received their first dose of acalabrutinib between 1 April 2020 and 1 April 2021.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Real-world progression free survival (rwPFS) | 12 months
  rwPFS will be defined as the time from index date until earliest record of real-world progression event as determined by physicians' assessment, or death (if no progression) or end of follow-up (for censored observations) whilst on first line treatment.
Real-world progression free survival (rwPFS) | 24 months
  rwPFS will be defined as the time from index date until earliest record of real-world progression event as determined by physicians' assessment, or death (if no progression) or end of follow-up (for censored observations) whilst on first line treatment.
Real-world progression free survival (rwPFS) | 36 months
  rwPFS will be defined as the time from index date until earliest record of real-world progression event as determined by physicians' assessment, or death (if no progression) or end of follow-up (for censored observations) whilst on first line treatment.
Real-world progression free survival (rwPFS) | 48 months
  rwPFS will be defined as the time from index date until earliest record of real-world progression event as determined by physicians' assessment, or death (if no progression) or end of follow-up (for censored observations) whilst on first line treatment.
Real-world progression free survival (rwPFS) | 60 months
  rwPFS will be defined as the time from index date until earliest record of real-world progression event as determined by physicians' assessment, or death (if no progression) or end of follow-up (for censored observations) whilst on first line treatment.

SECONDARY OUTCOMES:
Real-world overall survival (rwOS) | 12 months
  rwOS will be defined as the time from index date up to death or last date the patient was known to be alive (for censored observations).
Real-world overall survival (rwOS) | 24 months
  rwOS will be defined as the time from index date up to death or last date the patient was known to be alive (for censored observations).
Real-world overall survival (rwOS) | 36 months
  rwOS will be defined as the time from index date up to death or last date the patient was known to be alive (for censored observations).
Real-world overall survival (rwOS) | 48 months
  rwOS will be defined as the time from index date up to death or last date the patient was known to be alive (for censored observations).
Real-world overall survival (rwOS) | 60 months
  rwOS will be defined as the time from index date up to death or last date the patient was known to be alive (for censored observations).
Real-world response rate (rwRR) | 12 months
  rwRR will be defined as the proportion of patients with a recorded significant anti-cancer response and will be defined here as the sum of complete response, partial response and partial response + lymphocytosis. Response will be based on the on the documented assessment of the local investigator.
Real-world response rate (rwRR) | 24 months
  rwRR will be defined as the proportion of patients with a recorded significant anti-cancer response and will be defined here as the sum of complete response, partial response and partial response + lymphocytosis. Response will be based on the on the documented assessment of the local investigator.
Real-world response rate (rwRR) | 36 months
  rwRR will be defined as the proportion of patients with a recorded significant anti-cancer response and will be defined here as the sum of complete response, partial response and partial response + lymphocytosis. Response will be based on the on the documented assessment of the local investigator.
Real-world response rate (rwRR) | 48 months
  rwRR will be defined as the proportion of patients with a recorded significant anti-cancer response and will be defined here as the sum of complete response, partial response and partial response + lymphocytosis. Response will be based on the on the documented assessment of the local investigator.
Real-world response rate (rwRR) | 60 months
  rwRR will be defined as the proportion of patients with a recorded significant anti-cancer response and will be defined here as the sum of complete response, partial response and partial response + lymphocytosis. Response will be based on the on the documented assessment of the local investigator.
Real-world clinical progression free survival 2 (rwPFS2) | 12 months
  rwPFS2 will be defined as the time from index date to the date of the second record of real-world progression (as determined by physicians' assessment) or death due to any cause (if no progression), whichever occurs first whilst on second line treatment. If there is no second progression or the patient is lost to follow-up, PFS2 will be censored at the time of the last available tumour assessment.
Real-world clinical progression free survival 2 (rwPFS2) | 24 months
  rwPFS2 will be defined as the time from index date to the date of the second record of real-world progression (as determined by physicians' assessment) or death due to any cause (if no progression), whichever occurs first whilst on second line treatment. If there is no second progression or the patient is lost to follow-up, PFS2 will be censored at the time of the last available tumour assessment.
Real-world clinical progression free survival 2 (rwPFS2) | 36 months
  rwPFS2 will be defined as the time from index date to the date of the second record of real-world progression (as determined by physicians' assessment) or death due to any cause (if no progression), whichever occurs first whilst on second line treatment. If there is no second progression or the patient is lost to follow-up, PFS2 will be censored at the time of the last available tumour assessment.
Real-world clinical progression free survival 2 (rwPFS2) | 48 months
  rwPFS2 will be defined as the time from index date to the date of the second record of real-world progression (as determined by physicians' assessment) or death due to any cause (if no progression), whichever occurs first whilst on second line treatment. If there is no second progression or the patient is lost to follow-up, PFS2 will be censored at the time of the last available tumour assessment.
Real-world clinical progression free survival 2 (rwPFS2) | 60 months
  rwPFS2 will be defined as the time from index date to the date of the second record of real-world progression (as determined by physicians' assessment) or death due to any cause (if no progression), whichever occurs first whilst on second line treatment. If there is no second progression or the patient is lost to follow-up, PFS2 will be censored at the time of the last available tumour assessment.
Frequency of acalabrutinib dose interruptions | Through study completion, an average of 5 years
  A treatment interruption will be defined as clinician or patient-initiated temporary treatment cessation of acalabrutinib, where treatment is known to have been recommenced at any time within the observation window (without initiation on a different systemic treatment for CLL in the intervening period).

CONTACTS AND LOCATIONS:
Overall Officials: Toby A Eyre, Principal Investigator — Department of Clinical Haematology, Oxford University Hospitals NHS Foundation Trust, Oxford, UK
Locations (28):
- United Kingdom (28):
  - Research Site, Aylesbury
  - Research Site, Bath
  - Research Site, Birmingham
  - Research Site, Bournemouth
  - Research Site, Cardiff
  - Research Site, Cornwall
  - Research Site, Dartford
  - Research Site, Derby
  - Research Site, Doncaster
  - Research Site, Dorset
  - Research Site, Eastbourne
  - Research Site, Hull
  - Research Site, Leicester
  - Research Site, Lincoln
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Mid Yorkshire
  - Research Site, Middlesbrough
  - Research Site, Newcastle
  - Research Site, North Shields
  - Research Site, Norwich
  - Research Site, Nottingham
  - Research Site, Oxford
  - Research Site, Plymouth
  - Research Site, Southampton
  - Research Site, Stockton-on-Tees
  - Research Site, Stoke-on-Trent
  - Research Site, Wigan